CLINICAL TRIAL: NCT03377127
Title: PHARM-MD; An Open-Label, Randomized Controlled Phase II Study to Evaluate the Efficacy of a Pharmacist Managed Diabetes Clinic in High-Risk Diabetes Patients
Brief Title: Impact of Pharmacy Clinic on Diabetes Management
Acronym: PharmaMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Alexandra Halalau, Director of Internal Medicine Research, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-494
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; pharmacy clinic; education; diabetes complications; hemoglobin A1c; health-care cost; 'no show' rate; compliance; diabetes core measures
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Diabetes Complications; Patient Compliance | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a randomized open-label, controlled parallel group trial of a pharmacist managed diabetes clinic in high-risk diabetes patients, with a 1:1 allocation to either standard of care (SOC) or SOC and PMDC and a 6-month and 12-month follow-up.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patients and physicians will not be blinded to the intervention. However, the data collectors and the data analysts will be unaware of the patients allocation. The outcome assessors will also not be aware of the allocation. The biostatistician will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): The control group patients will be managed by their assigned PCPs, per Standard of Care (SOC), per American Diabetes Association Guidelines. Management per standard of care includes referrals to ophthalmology for dilated eye exam, nephrology for nephropathy management, cardiology for macrovascular complications management, neurology for neuropathy or neurologic complications, diabetic education, laboratory studies, and vaccinations and will be ordered or performed at the discretion of each patient's PCP
  Interventions: Other: Standard of Care (SOC)
- SOC and PMDC (Experimental): The intervention group patients will be managed by their assigned primary care physicians (PCPs), per American Diabetes Association Guidelines for Standard of Care (SOC) and will have scheduled six extra face-to-face visits with the pharmacists for the 6 month duration of the intervention. The pharmacy managed diabetes clinic (PMDC) visit encounters will focus on patient identified goals for the management of their diabetes. Pharmacists have the discretion to make medication adjustments and initiate new medications pertinent to the management of diabetic comorbidities. The model is a collaborative practice agreement between the pharmacist and the primary care physician.
  Interventions: Behavioral: Pharmacy Managed Diabetes Clinic (PMDC); Other: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: Pharmacy Managed Diabetes Clinic (PMDC) — The PMDC visit encounters will focus on patient identified goals for the management of their diabetes. Initial visit in the PMDC will be 60-90 minutes with follow up visits lasting 30-45 minutes.
  Arms: SOC and PMDC
Other: Standard of Care (SOC) — Standard of care will be delivered at the physician discretion per the current American Diabetes Association recommendations

SUMMARY:
The Beaumont Hospital Royal Oak Outpatient Clinic (and other listed Beaumont recruiting locations) care for over 900 patients with diabetes. In an effort to improve the care provided to our patients, a pharmacist managed diabetes clinic (PMDC) was created. The investigators looked at patients with high-risk diabetes who have received education in the PMDC and compared them to patients that didn't not receive the pharmacy education. Our preliminary data showed a significant decrease in Hemoglobin A1c in the PMDC compared to our standard care cohort. Hemoglobin A1c is a marker of the severity of diabetes mellitus. Based on this data, we designed a randomized controlled trial to better assess the impact of a PMDC on diabetic outcomes.

DETAILED DESCRIPTION:
Over the past 20 years, the number of adults with diabetes has tripled in the United States. According to the Centers for Disease Control (CDC), diabetes mellitus (DM) affected 30.2 million American adults in 2015.

Previous studies showed that for each 1% reduction in hemoglobin A1c (HbA1c), there was a corresponding 14% reduction in myocardial infarction, 12% reduction in stroke, and a 37% reduction of microvascular complications.

Based on our preliminary data, a Pharmacist Managed Diabetes Clinic (PMDC) had a decrease in HbA1c of 2.2% in the high-risk diabetes patients from the PMDC cohort versus 0.9% in the standard care cohort (p=0.006). At six months there was a decrease in HbA1c of 3.2% in the PMDC and 1.2% in the standard care cohort (p=0.044).

Our hypothesis is that a pharmacist managed diabetes clinic focused on patient identified diabetes management gaps and goals would have a significant positive impact on diabetes core measures and will result in a higher quality of care at a lower price. A randomized controlled trial (RCT) of our PMDC would provide further clarity on the impact on patient outcomes and important evidence with regard to how the physicians can deliver the best care for this high-risk population.

Trial design This is a randomized open-label, controlled parallel group trial of a pharmacist managed diabetes clinic in high-risk diabetes patients, with a 1:1 allocation to either standard of care (SOC) or SOC and PMDC and a 6-month and 12-month follow-up.

Methods:

The study will be conducted at the listed recruiting sites at Beaumont Hospital. Michigan. The outpatient clinic is a resident clinic that delivers medical care to over 920 patients with diabetes mellitus. The clinic is based on campus at Beaumont Hospital, Royal Oak. Potential subjects with high-risk diabetes mellitus will be identified through weekly reports and from the daily schedule and will be recruited from this pool of patients exclusively.

Intervention The patients will be enrolled over a 6-month period and will be randomly assigned to control group (usual care) and the intervention group (usual care plus PMDC visits). The PMDC is a pharmacist-led clinic that has been functioning in our outpatient clinic since January 2015 and is considered an available resource.

The intervention group patients will be managed by their assigned primary care physicians (PCPs), per standard of care and will have scheduled six extra face-to-face visits with the pharmacists for the 6 month duration of the intervention. The PMDC visits will be scheduled more frequent in the first 2 months of the intervention to ensure patients' engagement and provide enough opportunities and time to address all the patients' goals and concerns. The PMDC visit encounters will focus on patient identified goals for the management of their diabetes. Initial visit in the PMDC will be 60-90 minutes with follow up visits lasting 30-45 minutes. Patients will be asked to describe their own gaps in knowledge and to identify their own management goals. Identification of knowledge gaps will allow targeted patient education to close those gaps. Other educational opportunities will potentially include diabetes mellitus pathophysiology, blood glucose goals, HbA1c goals, management of hyperglycemic and hypoglycemic episodes, review of medications, and counseling regarding diet and exercise. Pharmacists have the discretion to make medication adjustments and initiate new medications pertinent to the management of diabetic comorbidities. The model is a collaborative practice agreement between the pharmacist and the primary care physician.

The control group patients will be managed by their assigned PCPs, per standard of care. Management per standard of care includes referrals to ophthalmology for dilated eye exam, nephrology for nephropathy management, cardiology for macrovascular complications management, neurology for neuropathy or neurologic complications, diabetic education, laboratory studies, and vaccinations and will be ordered or performed at the discretion of each patient's PCP.

Outside the intervention, the participants in both groups will be treated identical. They will participate in the standard of care visits at baseline, at 3 months and at 6 months. These visits (visit 1, 6 and 9 in the intervention group and visit 1, 2 and 3 in the standard of care group) will be provided by each patient's primary care physician

ELIGIBILITY:
Inclusion Criteria:

* high risk diabetes mellitus type 2 patients (hemoglobin ≥ 9%)
* not currently enrolled in PMDC.
* established with a primary care resident internal medicine or medicine-pediatrics resident.
* have a diagnosis of diabetes mellitus type 2.

Exclusion Criteria:

* Patients will be excluded if they have been seen by the PMDC within the past 3 months.
* under 18 years of age or over 75 years of age.
* documented as having type 1 diabetes or
* latent autoimmune diabetes of adults.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra I Halalau, MD, Principal Investigator — Director of Internal Medicine Research
Locations (4):
- United States (4):
  - Beaumont Geriatric Assessment Center, Berkley, Michigan
  - Beaumont Outpatient Clinic, Royal Oak, Michigan
  - Beaumont Internal Medicine Center, Southfield, Michigan
  - Norton, Klein, Hug, Sabin and Maddens Internal Medicine & Primary Care Practice, Troy, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halalau A, Sonmez M, Uddin A, Karabon P, Scherzer Z, Keeney S. Efficacy of a pharmacist-managed diabetes clinic in high-risk diabetes patients, a randomized controlled trial - "Pharm-MD" : Impact of clinical pharmacists in diabetes care. BMC Endocr Disord. 2022 Mar 16;22(1):69. doi: 10.1186/s12902-022-00983-y. PMID 35296307
- [Derived] Halalau A, Shelden D, Keeney S, Hehar J. Pharm-MD; an open-label, randomized controlled, phase II study to evaluate the efficacy of a pharmacist-managed diabetes clinic in high-risk diabetes patients - study protocol for a randomized controlled trial. Trials. 2018 Aug 24;19(1):458. doi: 10.1186/s13063-018-2836-8. PMID 30143033

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Of Care: The control group patients will be managed by their assigned PCPs, per Standard of Care (SOC), per American Diabetes Association Guidelines. Management per standard of care includes referrals to ophthalmology for dilated eye exam, nephrology for nephropathy management, cardiology for macrovascular complications management, neurology for neuropathy or neurologic complications, diabetic education, laboratory studies, and vaccinations and will be ordered or performed at the discretion of each patient's PCP
  Standard of Care (SOC): Standard of care will be delivered at the physician discretion per the current American Diabetes Association recommendations
Period: Overall Study
Arm/Group | Standard Of Care | SOC and PMDC
Started | 42 | 44
Completed | 42 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Of Care | SOC and PMDC | Total
Number analyzed (Participants) | 42 | 44 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.40 (8.10) | 52.00 (9.67) | 52.69 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 16 | 20 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 26 | 46
  White | 21 | 17 | 38
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 44 | 86

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c at 6 Months
Description: change from baseline in Hemoglobin A1c, measured in % DCCT (Diabetes Control and Complications Trial) units
Time Frame: 6 months
Population: Data missing for 15 subjects, did not complete assessment.
Measure: Mean (Standard Deviation); unit: percentage of DCCT units
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 34 | 37
percentage of DCCT units | -1.32 (1.66) | -2.85 (2.69)

2. Primary Outcome: Hemoglobin A1c at 12 Months
Description: change from baseline in Hemoglobin A1c
Time Frame: 12 months
Population: Data missing for 25 subjects, did not complete assessment.
Measure: Mean (Standard Deviation); unit: percentage of DCCT unit
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 31 | 30
percentage of DCCT unit | -1.52 (1.92) | -2.79 (2.41)

3. Secondary Outcome: Hemoglobin A1c Less Than 8% at 6 Months
Description: Percentage of patients achieving a hemoglobin A1c measurement of less than 8.0%
Time Frame: 6 months
Population: Data missing for 15 subjects, did not complete assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 34 | 37
Participants | 10 | 21

4. Secondary Outcome: Hemoglobin A1c Less Than 8% at 12 Months
Description: Percentage of patients achieving a hemoglobin A1c measurement of less than 8.0% DCCT units
Time Frame: 12 months
Population: Data missing for 25 subjects, did not complete assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 31 | 30
Participants | 11 | 16

5. Secondary Outcome: Change in Hemoglobin A1c From 6 to 12 Months
Description: The change in hemoglobin A1c (HbA1c), between 6 months and 12 months after randomization.
Time Frame: 12 months
Population: data were not collected or analyzed for this outcome for any participant
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Achievement of Annual Lipid Panel Testing
Description: percentage of patients complying with annual lipid testing
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 42 | 44
Participants | 24 | 26

7. Secondary Outcome: Statin Compliance
Description: Percentage of patients compliant with statin therapy per the 2013 American College of Cardiology / American Heart Association guidelines.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 42 | 44
Participants | 37 | 35

8. Secondary Outcome: Blood Pressure
Description: Percentage of patients achieving Blood pressure goal of less than 140/90 at the end of the trial period.
Time Frame: 12 months
Population: Data missing for 23 subjects, did not complete assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 31 | 32
Participants | 26 | 21

9. Secondary Outcome: Annual Retinopathy Examination
Description: Percentage of patients compliant with annual retinopathy examination
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 42 | 44
Participants | 25 | 25

10. Secondary Outcome: Annual Nephropathy Examination
Description: Percentage of patients compliant with annual nephropathy examination
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 42 | 44
Participants | 30 | 26

11. Secondary Outcome: Annual Neuropathy Examination
Description: Percentage of patients compliant with annual neuropathy examination
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 42 | 44
Participants | 30 | 29

12. Secondary Outcome: Annual Influenza Vaccine
Description: Percentage of patients compliant with annual influenza vaccine
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 42 | 44
Participants | 21 | 20

13. Secondary Outcome: Annual Pneumonia Vaccine
Description: Percentage of patients compliant with annual pneumonia vaccine
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 42 | 44
Participants | 31 | 27

14. Secondary Outcome: Quality of Life Assessment
Description: Difference between quality of life assessment via the World Health Organization BREF-Quality Of Life at baseline and 12 months.The WHOQOL-BREF consists of 4 domains, Physical Health, Psychological, Social Relationships, and Environment. Each domain is comprised of multiple questions that are considered together in the derivation of each domain score. In addition to the 4 domains, the WHOQOL-BREF includes two stand-alone questions to assess rated QOL and Satisfaction with Health questionnaire administered at baseline and at the conclusion of the trial period. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life) and range from a minimum of 4 to a maximum of 20. The mean score of items within each domain is used to calculate the domain score.A Likert scale from 1-7 was used. (1 - not affected, 7- extremely affected) We compared and reported the mean difference in between 6 months data and baseline data.
Time Frame: 12 months
Population: Data missing for 34 subjects, did not complete assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 29 | 23
score on a scale | -0.31 (2.05) | -0.78 (2.07)

15. Secondary Outcome: Diabetes Related EC Visits at 6 Months
Description: Number of Emergency Center (EC) visits related to hyperglycemia or hypoglycemia
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 42 | 44
number of visits | 0.10 (0.37) | 0.00 (0.00)

16. Secondary Outcome: Diabetes Related EC Visits at 12 Months
Description: Number of Emergency Center (EC) visits related to hyperglycemia or hypoglycemia
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 42 | 44
number of visits | 0.12 (0.40) | 0.02 (0.15)

17. Secondary Outcome: Total EC Visits at 6 Months
Description: Number of Emergency Center (EC) visits
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 42 | 44
number of visits | 0.62 (0.99) | 0.68 (1.12)

18. Secondary Outcome: Total EC Visits at 12 Months
Description: Number of Emergency Center (EC) visits
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 42 | 44
number of visits | 1.05 (1.29) | 1.09 (1.65)

19. Secondary Outcome: Inpatient Visits
Description: Total number of inpatient visits
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 42 | 44
number of visits | 0.71 (1.94) | 0.73 (1.13)

20. Secondary Outcome: Outpatient Visits
Description: total number of outpatient visits
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 42 | 44
number of visits | 7.60 (5.69) | 7.55 (4.25)

21. Secondary Outcome: No-show
Description: percentage of visits missed in clinic
Time Frame: 12 months
Population: data were not collected or analyzed for this outcome for any participant
Arm/Group | Standard Of Care | SOC and PMDC
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Standard Of Care | SOC and PMDC
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT03377127/Prot_SAP_002.pdf
  • Informed Consent Form (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT03377127/ICF_000.pdf